CLINICAL TRIAL: NCT01473134
Title: A Randomized Clinical Study to Compare the Safety and Efficacy of the Oxford Cementless Partial Knee System
Brief Title: Safety and Efficacy of the Oxford Cementless Partial Knee System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDE: G100123; ORTHO.CR.US30 (Other: Biomet)
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Avascular Necrosis of the Medial Femoral Condyle
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Oxford Cementless Partial Knee (Experimental): Oxford Partial Knee implanted without bone cement.
  Interventions: Device: Oxford Cementless Partial Knee
- Oxford Cemented Partial Knee (Active Comparator): Oxford Partial Knee applied with bone cement.
  Interventions: Device: Oxford Cemented Partial Knee

INTERVENTIONS:
Device: Oxford Cementless Partial Knee — Oxford Partial Knee applied without bone cement.
  Arms: Oxford Cementless Partial Knee
Device: Oxford Cemented Partial Knee — Oxford Partial Knee applied with bone cement.
  Arms: Oxford Cemented Partial Knee

SUMMARY:
The objective of this clinical investigation is to evaluate the safety and effectiveness of the Oxford® Cementless Partial Knee System. The Oxford® Cementless Partial Knee System is intended to help the patients diagnosed with osteoarthritis or avascular necrosis gain mobility and decrease pain. All of the risks common to a conventional joint replacement are possible with this device as certain risks are associated with any invasive procedures. The study is designed to document and compare the clinical and radiographic results of the Oxford® Cementless Partial Knee System to those of the cemented Oxford® Partial Knee System (control treatment).

DETAILED DESCRIPTION:
Prospectively controlled, randomized Investigational study. Patients are asked to come in pre-operatively, surgery, 6 weeks, 6 months, 1 year, 2 years and annually until the last patient reaches their 2 year visit. Product has not been cleared for use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a preoperative Knee Society Assessment Score of <70
* Patients undergoing primary partial knee arthroplasty as unilateral arthroplasty or bilateral arthroplasty, simultaneously or otherwise
* Patients diagnosed with osteoarthritis or avascular necrosis limited to the medial compartment of the operative knee joint
* Male or female patients who are at least 21 years of age at the time of surgery
* Patients with full thickness cartilage loss, with or without bone loss in the medial compartment
* Patients with functionally intact Anterior Cruciate Ligament (ACL) and Posterior Cruciate Ligament (PCL)
* Patients who needs to obtain relief of pain and/or improved function in their knee
* Patients with fixed flexion deformity <15 degrees
* Patients who are able to follow postoperative care instructions
* Patients who are willing and able to return for scheduled follow-up evaluations
* Patients in which natural alignment can be restored
* Patients who have completed a valid, Institutional Review Board (IRB) approved Informed Consent Form
* Patients with child-bearing potential who voluntarily agree to prevent pregnancy for 2 years following device implantation

Exclusion Criteria:

* Patients with a preoperative Knee Society Assessment Score of greater than or equal to 70
* Patients in which the device would be used to revise a failed prosthesis
* Patients who are less than 21 years of age, at the time of surgery
* Disease or damage to the lateral part of the knee that in the investigator's opinion contraindicates a partial knee replacement
* Patients diagnosed with rheumatoid arthritis or other forms of inflammatory joint disease
* Patients diagnosed with a failed upper tibial osteotomy in the operative knee
* Patients diagnosed with post-traumatic arthritis after tibial plateau fracture
* Patients who have had a patellectomy
* Patients with a flexion deformity > 15 degrees
* Patients with a fixed varus deformity > 15 degrees
* Patients who have rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Patients with a fused knee on operative side(s)
* Patients who have active or suspected infection, local or systemic that, in the opinion of the investigator, may put patients at undue risk
* Patients with pre-existing condition(s) that may interfere with the survival of the implants or their outcomes, including:

  * Sickle Cell Anemia
  * Lower extremity muscular atrophy
  * Neuromuscular disease
  * Vascular insufficiency
  * Metabolic Disorders which impair bone formation
  * Paget's Disease
  * Charcot's Disease
  * Osteomalacia
  * Severe Osteoporosis
* Patients with clinical conditions that may limit follow-up (in the opinion of the investigator) including:

  * Immunocompromised conditions (i.e. HIV)
  * Hepatitis
  * Tuberculosis
  * Neoplastic disease such as cancer of the prostate, lung, stomach, cervix, etc.
* Chronic renal failure
* Organ transplant (i.e. heart, liver, lung, etc.) recipients
* Known disease process that in the opinion of the investigator may limit long term (4 year) follow-up (i.e. multiple sclerosis, leukemia, lymphoma, etc.)
* Patients diagnosed with Parkinson's or Alzheimer's Disease
* Patients who have had an above-knee amputation in the contralateral leg
* Instability or deformity of the ligaments and/or surrounding soft tissue, which would preclude stability of the prostheses
* Patients with a known metal allergy
* Prisoners or, individuals who are known to be abusing drugs or alcohol or are mentally incompetent
* Patients who have received systemic steroids within the past 6 months or steroid injections into the affected knee within the previous 6 weeks prior to enrollment
* Patients who are pregnant
* Patients with severe valgus or varus knees (valgus or varus angulation of more than 20 degrees) where collateral ligament, iliotibial band, or popliteal release is required
* Patients who refuse to sign the IRB approved Informed Consent Form
* Participation in an interventional clinical research study procedure, other than a bilateral knee arthroplasty in this study, within the past 12 months
* Patients with a history of osteomyelitis or sepsis of the index knee
* Patients who require patellar resurfacing
* Patients who are not skeletally mature
* Patients who have had a total hip replacement procedure < 18 months prior to entering the study
* Patients who have had a contralateral non-study knee replacement procedure < 18 months prior to entering the study
* Patients who are found intraoperatively to have inadequate bone stock or other conditions that contraindicate a partial knee replacement

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (8):
- United States (8):
  - Orthopedic & Sports Medicine Center of Northern Indiana, Inc., Elkhart, Indiana
  - Midwest Center for Hip and Knee Surgery, Indianapolis, Indiana
  - Miller Orthopaedic Affiliates, Council Bluffs, Iowa
  - Twin City Orthopedics, Edina, Minnesota
  - OrthoCarolina, Huntersville, North Carolina
  - Joint Implant Surgeons, Inc, New Albany, Ohio
  - Texas Center for Joint Replacements, Plano, Texas
  - Anderson Orthopedic Clinic, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ELK1078R - bilateral subject was randomized to Investigational arm and received the Cementless device during the initial surgery. During the contralateral surgery, the cemented keel saw was used therefore, the Control device was implanted. Because this subject was randomized to Investigational and received 1 control knee, the investigational count in the participant flow is off by 1. A row was added with a note for this subject.
Units Other Than Participants: knees
Period: Overall Study
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Started | 207; 241 knees (ELK1078R - bilateral subject was randomized to Investigational arm and received the Cementless device during the initial surgery. During the contralateral surgery, the cemented keel saw was used therefore, the Control device was implanted according to the study protocol. Because this participant is in both the control and investigational groups it throws the 'participant' flow count off by 1. A row was added with the study completion reason "other" for this subject.) | 113; 137 knees
Completed | 152; 181 knees | 78; 95 knees
Not Completed | 55; 60 knees | 35; 42 knees
Not completed — Lost to Follow-up | 21 | 13
Not completed — Protocol Violation | 32 | 19
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 0 | 1
Not completed — ELK1078R: bilateral subject randomized to investigational, 2nd knee was cemented. | 1 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: knees
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee | Total
Number analyzed (Participants) | 207 | 113 | 320
Number analyzed (knees) | 241 | 137 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.7) | 66.4 (8.5) | 66.04 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 54 | 135
  Male | 126 | 59 | 185
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 207 | 113 | 320

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Success
Description: This is a binary endpoint in which a knee is either a "success" or "failure".
  To obtain a successful radiographic endpoint, a knee must meet the following criteria at the 22+ month interval.
  1. Absence of osteolysis
  2. No migration/subsidence of any femoral or tibial component
  3. Absence of fractured component
  Conversely, a radiographic failure is defined as follows:
  1. Presence of osteolysis defined as a radiolucency that is both progressive and is greater than 3 mm at its maximum interface in two or more contiguous zones OR a bony destructive lesion that is progressive in nature.
  2. Migration/subsidence of any femoral or tibial component defined as a component migration/subsidence of > 3 mm as compared to 6 week radiographs.
  3. A component fracture
Time Frame: 2 years
Population: The analysis was performed on the per protocol population who had a radiographic assessment at the 2+ year follow up interval. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees).
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 183 | 95
Number analyzed (knees) | 211 | 115
knees
  Successful | 198 | 112
  Failure | 13 | 3

2. Primary Outcome: Absence of Revision/Removal/Unanticipated Adverse Device Effect (UADE)
Description: This is a binary endpoint in which a knee is either a "success" or "failure". To obtain a successful result, a knee must reach the 2 year upper window limit with the device intact and without a component revision/removal or a UADE.
Time Frame: 2 Years
Population: The analysis was performed on the per protocol population who had an evaluation at the 2+ year follow up interval. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees).
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 186 | 101
Number analyzed (knees) | 216 | 122
knees
  Successful | 203 | 119
  Failures | 13 | 3

3. Primary Outcome: The Knee Society Assessment Score
Description: The Knee Society Assessment Score judges the parameters of pain, stability, and range of motion and flexion contracture, extension lag, and misalignment are deductions. The minimum score is 0 and maximum is 100, higher scores meaning a better outcome.
Time Frame: 2 Years
Population: The analysis was performed on the per protocol population who completed the The Knee Society Assessment Score at the 2+ year follow up interval.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 178 | 96
Number analyzed (Knees) | 204 | 116
score on a scale | 95.6 (8.3) | 95.5 (7.0)

4. Primary Outcome: The Knee Society Function Score
Description: The Knee Society Function Score considers walking distance and stair climbing, with deductions for walking aids. The minimum score is 0 and maximum is 100, higher scores meaning a better outcome.
Time Frame: 2 Year
Population: The analysis was performed on the per protocol population who completed the The Knee Society Function Score at the 2+ year follow up interval.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 179 | 100
Number analyzed (Knees) | 206 | 121
score on a scale | 89.4 (14.4) | 89.7 (14.1)

5. Secondary Outcome: Knee Society Assessment Score
Description: as for outcome 3
Time Frame: Pre-operation (baseline), 6 weeks, 6 months, and annually thereafter until study completion
Population: The analysis was performed on the per protocol population who completed the The Knee Society Assessment Score at each follow-up timepoint. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees). The "Overall Number of Participants Analyzed" is the number of study participants pre-operatively; the "Overall Number of Units Analyzed" refers to the number of knees with data available for analysis at each follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 207 | 114
Number analyzed (Knees) | 241 | 137
score on a scale
  Pre-op | 43.2 (11) | 45 (11)
  6 Week: number analyzed (Participants) | 206 | 110
  6 Week: number analyzed (Knees) | 239 | 133
  6 Week | 86.5 (13.7) | 87 (12.8)
  6 Month: number analyzed (Participants) | 194 | 103
  6 Month: number analyzed (Knees) | 223 | 121
  6 Month | 93.5 (10.3) | 94.2 (8.3)
  1 Year: number analyzed (Participants) | 184 | 96
  1 Year: number analyzed (Knees) | 210 | 114
  1 Year | 94.1 (9.5) | 95 (9.3)
  2 Year: number analyzed (Participants) | 171 | 92
  2 Year: number analyzed (Knees) | 194 | 112
  2 Year | 95.5 (8.5) | 95.6 (6.9)
  3 Year: number analyzed (Participants) | 142 | 68
  3 Year: number analyzed (Knees) | 162 | 81
  3 Year | 95.2 (8.7) | 94.4 (9.9)
  4 Year: number analyzed (Participants) | 98 | 46
  4 Year: number analyzed (Knees) | 107 | 52
  4 Year | 95.3 (8.6) | 94.2 (8.8)
  5 Year: number analyzed (Participants) | 60 | 28
  5 Year: number analyzed (Knees) | 65 | 34
  5 Year | 95 (9.1) | 94.4 (10.3)
  6 Year: number analyzed (Participants) | 27 | 13
  6 Year: number analyzed (Knees) | 30 | 14
  6 Year | 92.8 (13.3) | 93.6 (11.2)

6. Secondary Outcome: Knee Society Score Assessment for Bilateral Subjects
Description: as for outcome 3
Time Frame: Pre-operation (baseline), 6 weeks, 6 months, and annually thereafter until study completion
Population: The analysis was performed on the bilateral subjects in the per protocol population who had a Knee Society Assessment Score at each follow-up timepoint. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees). The "Overall Number of Participants Analyzed" is the number of study participants pre-operatively; the "Overall Number of Units Analyzed" refers to the number of knees with data available for analysis at each follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 50 | 27
Number analyzed (Knees) | 84 | 50
score on a scale
  Preop | 43.4 (10.7) | 46.0 (11.7)
  6 Week: number analyzed (Participants) | 50 | 25
  6 Week: number analyzed (Knees) | 83 | 48
  6 Week | 86.6 (14.5) | 87.7 (12.5)
  6 Month: number analyzed (Participants) | 48 | 23
  6 Month: number analyzed (Knees) | 77 | 41
  6 Month | 93.7 (10.9) | 95.6 (5)
  1 Year: number analyzed (Participants) | 48 | 21
  1 Year: number analyzed (Knees) | 74 | 39
  1 Year | 94.1 (8.6) | 95.3 (7.4)
  2 Year: number analyzed (Participants) | 45 | 23
  2 Year: number analyzed (Knees) | 68 | 43
  2 Year | 95.7 (8.6) | 95.4 (6.4)
  3 Year: number analyzed (Participants) | 39 | 19
  3 Year: number analyzed (Knees) | 59 | 32
  3 Year | 96.2 (6.1) | 92.5 (11.8)
  4 Year: number analyzed (Participants) | 34 | 9
  4 Year: number analyzed (Knees) | 43 | 15
  4 Year | 96.4 (6) | 92.9 (7.2)
  5 Year: number analyzed (Participants) | 15 | 7
  5 Year: number analyzed (Knees) | 20 | 13
  5 Year | 92.8 (13.3) | 92.8 (10)
  6 Year: number analyzed (Participants) | 6 | 1
  6 Year: number analyzed (Knees) | 9 | 2
  6 Year | 91.4 (9.9) | 100 (0)

7. Secondary Outcome: Knee Society Function Score at All Timepoints
Description: as for outcome 4
Time Frame: Pre-operation (baseline), 6 weeks, 6 months, and annually thereafter until study completion
Population: The analysis was performed on the per protocol population who completed the The Knee Society Assessment Score at each follow-up. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees). The "Overall Number of Participants Analyzed" is the number of study participants pre-operatively; the "Overall Number of Units Analyzed" refers to the number of knees with data available for analysis at each follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 207 | 114
Number analyzed (Knees) | 241 | 137
score on a scale
  Pre-op: number analyzed (Participants) | 207 | NA
  Pre-op | 58.1 (16) | 57.7 (17.7)
  6 Week: number analyzed (Participants) | 206 | 110
  6 Week: number analyzed (Knees) | 240 | 133
  6 Week | 65.4 (20.4) | 70.2 (18.5)
  6 Month: number analyzed (Participants) | 194 | 103
  6 Month: number analyzed (Knees) | 223 | 121
  6 Month | 86 (15.3) | 87.4 (15.2)
  1 Year: number analyzed (Participants) | 184 | 96
  1 Year: number analyzed (Knees) | 210 | 114
  1 Year | 87.9 (15.9) | 88 (15.4)
  2 Year: number analyzed (Participants) | 171 | 95
  2 Year: number analyzed (Knees) | 195 | 116
  2 Year | 89.9 (13) | 89.8 (14)
  3 Year: number analyzed (Participants) | 145 | 71
  3 Year: number analyzed (Knees) | 165 | 84
  3 Year | 88.5 (15) | 88.9 (12.8)
  4 Year: number analyzed (Participants) | 99 | 48
  4 Year: number analyzed (Knees) | 108 | 55
  4 Year | 87.1 (17.1) | 90 (11.1)
  5 Year: number analyzed (Participants) | 61 | 28
  5 Year: number analyzed (Knees) | 66 | 34
  5 Year | 86.7 (17.4) | 85.6 (15.2)
  6 Year: number analyzed (Participants) | 27 | 13
  6 Year: number analyzed (Knees) | 30 | 14
  6 Year | 83.2 (19.7) | 85.7 (17.9)

8. Secondary Outcome: Knee Society Function Score for Bilateral Subjects
Description: as for outcome 4
Time Frame: Pre-operation (baseline), 6 weeks, 6 months, and annually thereafter until study completion
Population: The analysis was performed on the bilateral subjects in the per protocol population who had a Knee Society Function Score at each follow-up timepoint. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees). The "Overall Number of Participants Analyzed" is the number of study participants pre-operatively; the "Overall Number of Units Analyzed" refers to the number of knees with data available for analysis at each follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 50 | 26
Number analyzed (Knees) | 84 | 50
score on a scale
  Pre-op | 60.1 (15.8) | 56.3 (19.3)
  6 Week: number analyzed (Participants) | 50 | 25
  6 Week: number analyzed (Knees) | 84 | 48
  6 Week | 65.8 (20.3) | 72 (15.3)
  6 Month: number analyzed (Participants) | 48 | 23
  6 Month: number analyzed (Knees) | 77 | 41
  6 Month | 84.5 (16) | 88.8 (14.7)
  1 Year: number analyzed (Participants) | 48 | 21
  1 Year: number analyzed (Knees) | 74 | 39
  1 Year | 85.3 (16.5) | 86.8 (16.1)
  2 Year: number analyzed (Participants) | 45 | 24
  2 Year: number analyzed (Knees) | 69 | 45
  2 Year | 88.6 (13) | 92.4 (10.5)
  3 Year: number analyzed (Participants) | 41 | 20
  3 Year: number analyzed (Knees) | 61 | 33
  3 Year | 89.3 (14.8) | 93.3 (8.4)
  4 Year: number analyzed (Participants) | 34 | 11
  4 Year: number analyzed (Knees) | 43 | 18
  4 Year | 90.7 (13.2) | 96.1 (6.1)
  5 Year: number analyzed (Participants) | 15 | 7
  5 Year: number analyzed (Knees) | 20 | 13
  5 Year | 90 (10.3) | 90.8 (13.2)
  6 Year: number analyzed (Participants) | 6 | 1
  6 Year: number analyzed (Knees) | 9 | 2
  6 Year | 82.2 (18.6) | 100 (0)
  7 Year: number analyzed (Participants) | 1 | 0
  7 Year: number analyzed (Knees) | 1 | 0
  7 Year | 60 (0) |

9. Secondary Outcome: Oxford Knee Score
Description: * 12-item self-report measure containing questions regarding the patient's pain and level of function
  * The scoring system ranges from 0-4 on each question with 4 representing maximum function and 0 representing poorest function.
  * Using this scale, the lowest, worst score is a 0, and the highest, best score is 48.
  * The OKS has 2 subscales:
    1. Pain
    2. Function The pain component score (OKS-PCS) consists of items 2, 3, 7, 11 and 12, and the functional component score consists of items 1, 4, 5, 6, 8, 9, and 10.
Time Frame: Pre-operation (baseline), 6 weeks, 6 months, and annually thereafter until study completion
Population: The analysis was performed on the per protocol population who completed the Oxford Knee Score at each follow-up timepoint. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees). The "Overall Number of Participants Analyzed" is the number of study participants pre-operatively; the "Overall Number of Units Analyzed" refers to the number of knees with data available for analysis at each follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 207 | 113
Number analyzed (Knees) | 241 | 137
score on a scale
  Pre-op | 23.7 (8.1) | 24.9 (7.6)
  6 Week: number analyzed (Participants) | 204 | 109
  6 Week: number analyzed (Knees) | 237 | 132
  6 Week | 32.4 (7.8) | 34.5 (7)
  6 Month: number analyzed (Participants) | 194 | 104
  6 Month: number analyzed (Knees) | 222 | 122
  6 Month | 41.8 (5.8) | 42.4 (6.1)
  1 Year: number analyzed (Participants) | 182 | 96
  1 Year: number analyzed (Knees) | 207 | 114
  1 Year | 42.9 (6.3) | 43.5 (5.7)
  2 Year: number analyzed (Participants) | 170 | 95
  2 Year: number analyzed (Knees) | 194 | 116
  2 Year | 44.5 (4.5) | 44.9 (3.9)
  3 Year: number analyzed (Participants) | 145 | 70
  3 Year: number analyzed (Knees) | 165 | 83
  3 Year | 44.6 (7.7) | 44.6 (6.2)
  4 Year: number analyzed (Participants) | 98 | 47
  4 Year: number analyzed (Knees) | 107 | 54
  4 Year | 44.3 (5.3) | 45 (5.9)
  5 Year: number analyzed (Participants) | 60 | 28
  5 Year: number analyzed (Knees) | 65 | 34
  5 Year | 43.7 (5.9) | 45.3 (4.9)
  6 Year: number analyzed (Participants) | 27 | 13
  6 Year: number analyzed (Knees) | 30 | 13
  6 Year | 41.3 (8.5) | 44.1 (7.1)
  7 Year: number analyzed (Participants) | 1 | 0
  7 Year: number analyzed (Knees) | 1 | 0
  7 Year | 44 (0) |

10. Secondary Outcome: Number of Knees Which Met the Criteria for Radiographic Success
Description: as for outcome 1
Time Frame: Pre-operation (baseline), 6 weeks, 6 months, 1y, 3y, 4y, 5y, 6y, 7y
Population: The analysis was performed on the per protocol population had a radiographic assessment at each follow-up timepoint. The analysis is at the knee level, not participant level (bilateral participants included as two individual knees). The "Overall Number of Participants Analyzed" is the number of study participants at 6 weeks; the "Overall Number of Units Analyzed" refers to the number of knees with data available for analysis at each follow-up timepoint.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 203 | 106
Number analyzed (Knees) | 235 | 129
Knees
  6 Week | 235 | 129
  6 Month: number analyzed (Participants) | 182 | 98
  6 Month: number analyzed (Knees) | 208 | 115
  6 Month | 208 | 115
  1 Year: number analyzed (Participants) | 184 | 96
  1 Year: number analyzed (Knees) | 208 | 113
  1 Year | 208 | 113
  2 Year: number analyzed (Participants) | 169 | 88
  2 Year: number analyzed (Knees) | 193 | 106
  2 Year | 180 | 103
  3 Year: number analyzed (Participants) | 129 | 66
  3 Year: number analyzed (Knees) | 147 | 79
  3 Year | 147 | 79
  4 Year: number analyzed (Participants) | 90 | 44
  4 Year: number analyzed (Knees) | 99 | 49
  4 Year | 99 | 49
  5 Year: number analyzed (Participants) | 58 | 27
  5 Year: number analyzed (Knees) | 63 | 32
  5 Year | 63 | 32
  6 Year: number analyzed (Participants) | 20 | 13
  6 Year: number analyzed (Knees) | 23 | 14
  6 Year | 23 | 14
  7 Year: number analyzed (Participants) | 1 | 0
  7 Year: number analyzed (Knees) | 1 | 0
  7 Year | 1 |

11. Secondary Outcome: Patient Assessment of Satisfaction
Description: At each postoperative assessment using the Analysis Windows, patients were asked to indicate their level of satisfaction with the operated knee. The potential outcomes were Very Satisfied, Satisfied, Uncertain and Unsatisfied.
Time Frame: 6 weeks, 6 months, and annually thereafter until study completion
Population: This analysis is done at the knee-level, not participant level. Bilateral participants were allowed in the study. The "Overall Number of Participants Analyzed" is the number of study subjects analyzed (some with unilateral and some with bilateral knees); the "Overall Number of Units Analyzed" refers to the number of knees analzyed. Also, not every participant returned for every follow-up visit. The "Number Analyzed" in each row/visit below shows the number of knees analyzed at each follow-up.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
Number analyzed (Participants) | 204 | 109
Number analyzed (Knees) | 237 | 132
Knees
  6 Week: Very Satisfied | 151 | 95
  6 Week: Satisfied | 60 | 27
  6 Week: Uncertain | 23 | 9
  6 Week: Unsatisfied | 3 | 1
  6 Month: number analyzed (Participants) | 194 | 105
  6 Month: number analyzed (Knees) | 222 | 123
  6 Month: Very Satisfied | 166 | 95
  6 Month: Satisfied | 35 | 20
  6 Month: Uncertain | 19 | 5
  6 Month: Unsatisfied | 2 | 3
  1 Year: number analyzed (Participants) | 179 | 96
  1 Year: number analyzed (Knees) | 204 | 114
  1 Year: Very Satisfied | 156 | 93
  1 Year: Satisfied | 38 | 17
  1 Year: Uncertain | 8 | 3
  1 Year: Unsatisfied | 2 | 1
  2 Years: number analyzed (Participants) | 170 | 95
  2 Years: number analyzed (Knees) | 194 | 116
  2 Years: Very Satisfied | 158 | 100
  2 Years: Satisfied | 27 | 12
  2 Years: Uncertain | 8 | 3
  2 Years: Unsatisfied | 1 | 1
  3 Years: number analyzed (Participants) | 145 | 70
  3 Years: number analyzed (Knees) | 165 | 83
  3 Years: Very Satisfied | 143 | 76
  3 Years: Satisfied | 17 | 3
  3 Years: Uncertain | 4 | 3
  3 Years: Unsatisfied | 1 | 1
  4 Years: number analyzed (Participants) | 98 | 47
  4 Years: number analyzed (Knees) | 107 | 54
  4 Years: Very Satisfied | 89 | 51
  4 Years: Satisfied | 16 | 1
  4 Years: Uncertain | 2 | 2
  4 Years: Unsatisfied | 0 | 0
  5 Years: number analyzed (Participants) | 60 | 28
  5 Years: number analyzed (Knees) | 65 | 34
  5 Years: Very Satisfied | 53 | 32
  5 Years: Satisfied | 8 | 0
  5 Years: Uncertain | 3 | 2
  5 Years: Unsatisfied | 1 | 0
  6 Years: number analyzed (Participants) | 27 | 13
  6 Years: number analyzed (Knees) | 30 | 14
  6 Years: Very Satisfied | 24 | 13
  6 Years: Satisfied | 4 | 0
  6 Years: Uncertain | 2 | 0
  6 Years: Unsatisfied | 0 | 1
  7 Years: number analyzed (Participants) | 1 | 0
  7 Years: number analyzed (Knees) | 1 | 0
  7 Years: Very Satisfied | 1 |
  7 Years: Satisfied | 0 |
  7 Years: Uncertain | 0 |
  7 Years: Unsatisfied | 0 |

ADVERSE EVENTS:
Time Frame: AEs were collected from post-op until study completion (up to 7 years for the longest-enrolled participants).
Description: Adverse Event Case Report Form (worksheet)
Arm/Group | Oxford Cementless Partial Knee | Oxford Cemented Partial Knee
All-Cause Mortality (participants affected / at risk) | 3/207 | 9/114
Serious Adverse Events (participants affected / at risk) | 17/207 | 10/114
Other Adverse Events (participants affected / at risk) | 114/207 | 53/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxford Cementless Partial Knee (N=207) | Oxford Cemented Partial Knee (N=114)
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Bearing Dislocation/Disassociation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Cellulitis/Redness/Blistering (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Deep Wound Infection (Infections and infestations) | 1 (1) | 0
Effusion/Swelling/Edema (Musculoskeletal and connective tissue disorders) | 2 (2) | 0
Femoral Implant Loosening (Injury, poisoning and procedural complications) | 1 (1) | 0
Hemarthrosis/Hemarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Hematoma (Vascular disorders) | 2 (2) | 0
Loose body and/or Osteophyte Removal (Surgical and medical procedures) | 0 | 1 (1)
Other Ipsilateral Knee Related Adverse Event (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Pain (progressive/persistent) (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Progressive Disease in Contralateral Compartment (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Subsidence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibial Fracture (Injury, poisoning and procedural complications) | 4 (4) | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxford Cementless Partial Knee (N=207) | Oxford Cemented Partial Knee (N=114)
Clicking/Popping/Crepitus/Grinding (Musculoskeletal and connective tissue disorders) | 13 (15) | 4 (4)
Effusion/Swelling/Edema (Musculoskeletal and connective tissue disorders) | 29 (33) | 9 (11)
Other Ipsilateral Knee Related Adverse Event (Injury, poisoning and procedural complications) | 36 (45) | 18 (27)
Pain (progressive/persistent) (General disorders) | 50 (63) | 22 (30)
Traumatic Injury (Study Knee) (Injury, poisoning and procedural complications) | 16 (21) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each participating PI has signed a Clinical Trial Agreement and results are not publicly available until FDA provides approval/closure of the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT01473134/Prot_SAP_000.pdf